CLINICAL TRIAL: NCT01535950
Title: A Multicenter, Randomized, Sham-controlled, Repeat-dose Study to Assess the Safety, Tolerability, Serum Pharmacokinetics, and Efficacy of Intravitreal LFG316 in Patients With Neovascular Age-related Macular Degeneration
Brief Title: Safety and Efficacy of Intravitreal LFG316 in Wet Age Related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLFG316A2202
Record Dates: First submitted 2012-02-10; First posted 2012-02-20 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2016-03

CONDITIONS: Neovascular Age-elated Macular Degeneration (Wet AMD); Exudative Macular Degeneration
Keywords: Age-related macular degeneration; intravitreal, neovascular; anti-vascular endothelial growth factor; wet AMD; Age-related; Macular degeneration; Intravitreal; Neovascular
MeSH Terms: conditions — Wet Macular Degeneration; Macular Degeneration

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- LFG316 (Experimental)
  Interventions: Drug: LFG316
- Sham (Sham Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LFG316
  Arms: LFG316
Drug: Placebo — Placebo will be administered as sham injections. Sham injections will involve placement of the syringe hub against the sclera, without use of a needle.
  Arms: Sham

SUMMARY:
This study will assess the safety and efficacy of LFG316 in patients with age related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Best corrected visual acuity (ETDRS scale) of 60 letters or less in the study eye.
* An active choroidal neovascular membrane attributable to neovascular AMD in at least one eye.
* History of treatment (at any time) with at least 3 doses of anti-VEGF therapy in the study eye.

Exclusion Criteria:

* History of recurrent non-response to anti-VEGF therapy in the study eye.
* In the study eye, retinal disease other than AMD (benign conditions of the vitreous and peripheral retina are not exclusionary).
* Choroidal neovascularization due to a cause other than AMD.
* In the study eye, media opacity that, in the investigator's opinion, could interfere with conduct of the study.
* History of infectious uveitis or endophthalmitis in either eye.
* Any of the following treatments to the study eye within 28 days prior to dosing: ranibizumab, bevacizumab, pegaptanib or other VEGF inhibitor.
* Any of the following within 90 days prior to dosing: photodynamic therapy or laser photocoagulation in the study eye; intravitreal steroid in the study eye; or intraocular surgery (including cataract surgery) in the study eye

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Number of anti-Vascular Endothelial Growth Factor (anti-VEGF) retreatments vs time | Day 1 to 113
  Number or retreatments with anti-VEGF treatments will be recorded

SECONDARY OUTCOMES:
The proportion of patients in the study that requires at least one treatment of anti-VEGF medication. | Day 1 and 113
  Number or retreatments with anti-VEGF treatments will be recorded
Effect of LFG316 on visual acuity | Day 1 and 113
  Early Treatment Diabetic Retinopathy Study" (ETDRS best corrected visual acuity measured under ESTDRS conditions Number of letters correctly read will be recorded.
Effect of LFG316 on central retinal thickness and choroidal neovascular membrane area, and drusen area/volume where applicable | Day 1 , Day 85 and Day 113 (starting from the day of first IVT injection until end of study)
  Summary statistics of these variables will be provided by treatment and visit/time. Treatment effect will be assessed by comparison of mean change from baseline to Day 85.
Serum concentrations of total LFG316 versus time | Days 1, 8, 15, 29, 43, 57, 71, 85 and 113
  Blood samples will be collected
Number of patients with adverse events | Day 113
  Adverse events will be determined based on descriptive analyses of vital signs, electrocardiogram (ECG) evaluation, and clinical safety laboratory evaluations. All abnormalities will be flagged and summary statistics will be provided by treatment and visit/time.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- United States (7):
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Torrance, California
  - Novartis Investigative Site, Fort Myers, Florida
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, West Columbia, South Carolina
  - Novartis Investigative Site, Abilene, Texas
  - Novartis Investigative Site, Fort Worth, Texas

REFERENCES:
- See also: Results for CLFG316A2202 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=12244